CLINICAL TRIAL: NCT00460122
Title: Pilot Study of the Incidence of HLA Class I and Class II Antibodies in Platelet Donors and Their Effects on the Transfusion Recipient
Brief Title: Effects of Antibodies to White Blood Cells on Platelet Transfusion Patients
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070125; 07-CC-0125
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2012-08-10

CONDITIONS: Healthy; Transfusion Reactions
Keywords: Human Leukocyte Antigens (HLA); Transfusion Reactions; Platelet Donors
MeSH Terms: conditions — Transfusion Reaction

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will determine if transfusion of platelets containing HLA antibodies (certain antibodies to white blood cells) are more likely to cause transfusion reactions than transfusion of platelets that do not contain HLA antibodies.

People 18 years of age or older who donate platelets at the NIH Clinical Center may be eligible for this study.

An extra tube of blood (about one teaspoon) is obtained from participating donors at the time of their donation at the NIH Platelet Center. The blood plasma in the extra tube is tested for HLA antibodies and antibodies to certain white blood cells called granulocytes. The research sample is assigned a code number for identification and sent to the HLA Laboratory in the Department of Transfusion Medicine.

DETAILED DESCRIPTION:
Leukocyte antibodies can cause febrile transfusion reactions, pulmonary reactions to granulocyte transfusions, and transfusion related acute lung injury (TRALI). Despite the fact that the role of leukocyte antibodies in these reactions was first described almost 50 years ago, and that TRALI is now the leading cause of transfusion related fatalities, much remains uncertain concerning the role of HLA antibodies in these reactions. The primary purpose of this study is to retrospectively and prospectively determine if the incidence and nature of transfusion reactions differs in Clinical Center (CC) patients that were transfused with platelet components from donors with HLA antibodies and those without HLA antibodies. In addition, this study will prospectively determine the incidence of HLA antibodies in the NIH Department of Transfusion Medicine (DTM) platelet donor population. In this natural history study a 10-mL blood sample will be drawn from 600 platelet donors at the time that they are in the DTM donating platelets and it will be tested for HLA antibodies in the DTM. The blood sample for HLA antibody testing will be collected with other samples collected as part of the regular platelet donation process. Reactions in platelet transfusion recipients will be assessed by reviewing CC and DTM patient records.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Both male and female donors
  2. Any ethnic group
  3. 18 years of age or older
  4. Must meet the criteria for donating platelets in the DTM

EXCLUSION CRITERIA:

1. Donors are not eligible to donate platelets in the DTM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2007-04-10; Study Completion 2012-08-10

CONTACTS AND LOCATIONS:
Overall Officials: David F Stroncek, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Toy P, Popovsky MA, Abraham E, Ambruso DR, Holness LG, Kopko PM, McFarland JG, Nathens AB, Silliman CC, Stroncek D; National Heart, Lung and Blood Institute Working Group on TRALI. Transfusion-related acute lung injury: definition and review. Crit Care Med. 2005 Apr;33(4):721-6. doi: 10.1097/01.ccm.0000159849.94750.51. PMID 15818095
- [Background] Goldman M, Webert KE, Arnold DM, Freedman J, Hannon J, Blajchman MA; TRALI Consensus Panel. Proceedings of a consensus conference: towards an understanding of TRALI. Transfus Med Rev. 2005 Jan;19(1):2-31. doi: 10.1016/j.tmrv.2004.10.001. PMID 15830325
- [Background] BRITTINGHAM TE. Immunologic studies on leukocytes. Vox Sang. 1957 Sep;2(4):242-8. doi: 10.1111/j.1423-0410.1957.tb03699.x. No abstract available. PMID 13496693